CLINICAL TRIAL: NCT00957749
Title: A Multicenter, Open-Label Study of the Safety, Tolerability, and Pharmacodynamics of Intravenously Administered cPMP (Precursor Z) in Patients With Molybdenum Cofactor Deficiency Type A
Brief Title: Study of cPMP (Precusor Z) to Treat Molybdenum Cofactor Deficiency (MoCD) Type A
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: IND application was withdrawn, and therefore study listing is being withdrawn.
Sponsor: Orphatech Pharmaceuticals, GmbH (Industry)
Responsible Party: Robert Gianello, Orphatech GmbH
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cPMP01-08
Record Dates: First submitted 2009-07-10; First posted 2009-08-12 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Molybdenum Cofactor Deficiency Type A
MeSH Terms: conditions — Molybdenum Cofactor Deficiency, Complementation Group A | interventions — nulibry; molybdopterin synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cPMP (Experimental)
  Interventions: Drug: cPMP

INTERVENTIONS:
Drug: cPMP — Intravenous solution administered daily. Dose titrated from 80 μg/kg on Days 1-12 to 120 μg/kg on Days 13-34 to 160 μg/kg for days 35-90.
  Other Names: Cyclic pyranopterin monophosphate; Precursor Z

SUMMARY:
Molybdenum Cofactor Deficiency Type A (MoCD) is a very rare autosomal recessive disorder that is essentially fatal early in life. Naturally occurring cPMP is present in the body of all healthy normal individuals. It is processed to molybdopterin, which is further processed to molybdenum cofactor. Molybdenum cofactor is essential for the function of important enzymes.

There is currently no treatment for MoCD, and affected infants develop severe neurological damage which often results in infant death.

This study is the first clinical trial to investigate the potential of replacement of cPMP to infants with MoCD Type A. The safety, tolerability, and pharmacodynamics of daily intravenous administration of cPMP over 3 months will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Neonate or infant, less then 6 weeks at the time of diagnosis, age less than 8 weeks at start of treatment with the study medication. It is important to diagnose the condition and initiate treatment as soon after birth as possible.
* Documented diagnosis of molybdenum cofactor deficiency (MoCD) Type A based on the absence of cPMP and the presence of sulfite and s-sulfocysteine in the urine, absence of urothione in the urine and genetic analysis showing a mutation in the MOCS1 gene
* A parent or legal guardian voluntarily provided written informed consent to participate in the study and comply with study procedures.
* Approval of the study protocol by the local HE / IRB and government or regulatory authorities (if applicable)

Exclusion Criteria:

* MoCD Type B (MOCS2 mutation) or Type C (gephyrin gene mutation)
* Sulfite oxidase deficiency
* Patients older than 6 weeks at the time of diagnosis

Max Age: 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Urine biomarkers SSC and sulfite | Daily collection throughout study; analyzed at 3 months

SECONDARY OUTCOMES:
neurological examination | collected daily; analyzed at 3 months
Safety measures (vital signs, adverse events) | collected daily; analyzed at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alex Veldman, MD, Principal Investigator — Monash Medical Centre
Locations (1):
- Monash Medical Centre, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Schwarz G, Santamaria-Araujo JA, Wolf S, Lee HJ, Adham IM, Grone HJ, Schwegler H, Sass JO, Otte T, Hanzelmann P, Mendel RR, Engel W, Reiss J. Rescue of lethal molybdenum cofactor deficiency by a biosynthetic precursor from Escherichia coli. Hum Mol Genet. 2004 Jun 15;13(12):1249-55. doi: 10.1093/hmg/ddh136. Epub 2004 Apr 28. PMID 15115759